CLINICAL TRIAL: NCT06077695
Title: Cognitive Remediation of Working Memory After Moderate to Severe Head Trauma. a SCED Study.
Brief Title: Cognitive Remediation of Working Memory Post Head Trauma
Acronym: Meta-SCED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RC31/22/0502
Record Dates: First submitted 2023-10-04; First posted 2023-10-11 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Head Trauma
Keywords: working memory; cognitive remediation; transcranial direct current stimulation
MeSH Terms: conditions — Craniocerebral Trauma | interventions — Transcranial Direct Current Stimulation; Cognitive Remediation

STUDY DESIGN:
Intervention Model Description: Single Case Experimental Design : SCEDs evaluate the effectiveness of an intervention by recruiting a small number of individuals (typically between 1 and 3). They are different from single case studies (or case reports). SCEDs are based on repeated measurements, sequential introduction of the intervention and specific visual and statistical methods of analyzing the results. The strength of SCED lies in the large number of repeated measurements and not in the number of subjects included.
Who Masked: Investigator
Masking Description: Repeated measurements, control measurements and neuropsychological examinations will be carried out by an examiner blinded to the intervention phase. The rehabilitator will not carry out these assessments. A neuropsychologist from the neuropsychology unit, not involved in the design and conduct of the Meta-SCED study, will carry out these examinations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 4 weeks phase A arm (Experimental): Phase A = Randomised duration of this phase : 4 weeks. each therapeutic therapeutic education sessions last 90 minutes.
  Phase B = therapeutic education with tDCS for 4 weeks
  Phase C = Cognitive remediation with tDCS for 4 weeks : Eight specific working memory remediation sessions will be carried out. These will be provided by a neuropsychologist. All cognitive remediation sessions will be individual, biweekly, lasting 1 hour 10 minutes for 4 weeks, for a total duration of 9 hours 20 minutes.
  Phase D = follow-up
  Interventions: Other: therapeutic education; Other: tDCS; Other: cognitive remediation
- 5 weeks phase A arm (Experimental): Phase A = therapeutic education. Randomised duration of this phase : 5 weeks. each therapeutic therapeutic education sessions last 90 minutes.
  Phase B = therapeutic education with tDCS for 4 weeks
  Phase C = Cognitive remediation with tDCS for 4 weeks : Eight specific working memory remediation sessions will be carried out. These will be provided by a neuropsychologist. All cognitive remediation sessions will be individual, biweekly, lasting 1 hour 10 minutes for 4 weeks, for a total duration of 9 hours 20 minutes.
  Phase D = follow-up
  Interventions: Other: therapeutic education; Other: tDCS; Other: cognitive remediation
- 6 weeks phase A arm (Experimental): Phase A = therapeutic education. Randomised duration of this phase : 6 weeks. each therapeutic therapeutic education sessions last 90 minutes.
  Phase B = therapeutic education with tDCS for 4 weeks
  Phase C = Cognitive remediation with tDCS for 4 weeks : Eight specific working memory remediation sessions will be carried out. These will be provided by a neuropsychologist. All cognitive remediation sessions will be individual, biweekly, lasting 1 hour 10 minutes for 4 weeks, for a total duration of 9 hours 20 minutes.
  Phase D = follow-up
  Interventions: Other: therapeutic education; Other: tDCS; Other: cognitive remediation

INTERVENTIONS:
Other: therapeutic education — The themes covered concern head trauma in the chronic phase.
Other: tDCS — The constant electric current will be delivered at an intensity of 2 mA for 20 minutes.The anode will be placed opposite the dorsolateral prefrontal area on the right. The cathode (or reference electrode) will be positioned opposite the supraorbital area on the left. This methodology is based on the general directions and results from scientific studies which aimed to improve the efficiency of neural networks engaged in attentional processes and working memory.
Other: cognitive remediation — Personalized sessions combining 2 approaches:•Retraining deficit components of working memory.exercise the strengthening of metacognition and the learning of "reorganization-facilitation" strategies. At the end of each exercise, the participant will be asked to analyze their performance and will benefit from feedback from the rehabilitator as well as a discussion on the use of the strategies. Finally, all of the proposed tasks will be made up of several levels of complexity; moving to a more complex stage will require more than 90% success in the exercise.•More ecological exercises will also be carried out in order to get as close as possible to the difficulties encountered by the patient on a daily basis. The examiner will guide the rehabilitation and propose tasks imitating his daily life.

SUMMARY:
Patients with working memory deficits due to a moderate to severe head injury will undergo a 5 month protocol including cognitive remediation with numerous exercises, transcranial direct current stimulation (tDCS), and therapeutic education.

DETAILED DESCRIPTION:
This study is a multiple baseline Single Case Experimental Design (SCED) across 3 patients and 2 behaviors (working memory performance, application of compensatory strategies).

The remediation program will include 4 intervention phases, and include patients with moderate or severe head trauma and expressing a cognitive complaint of working memory during the neuropsychological screening examination.

These patients will benefit from a neuropsychological assessment at inclusion then cognitive remediation treatment consisting of 4 phases. The duration of the baseline will be randomized. At the end of phases C and D, a new neuropsychological examination will be carried out.

Patients will have to come twice a week, for 12 weeks. All sessions will be individual.

* Phase A: Therapeutic education (Weeks 1 to 4) This first phase will include therapeutic education sessions lasting 90 minutes. The themes covered will concern Head trauma in the chronic phase. Cognitive and behavioral disorders secondary to traumatic brain injury (TBI) will not be addressed. The duration of this phase will be randomized.
* Phase B: tDCS + therapeutic education (Weeks 5 to 8) During this intervention phase, at each visit patients will have 20 minutes of tDCS stimulation and 70 minutes of therapeutic education.

Concerning tDCS stimulation, an electrical current of 2mA will be delivered using the electrodes for 20 min. The content of the therapeutic education sessions will be developed in the same way as for phase A.

• Phase C: tDCS + cognitive remediation (Weeks 9 to 12) During this intervention phase, at each visit, patients will have 20 minutes of tDCS stimulation and 70 minutes of specific cognitive remediation of working memory.

The cognitive remediation program will combine working memory retraining using computerized and paper-and-pencil supports as well as more ecological exercises that respond precisely to the difficulties encountered by the patient in daily life.

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe head trauma, defined by an initial Glasgow score ≤ 12/15, duration of post-traumatic amnesia superior to 24 hours and/or the presence of abnormalities on brain imaging,
* Moderate or severe head trauma occurring within a period greater than or equal to 3 months,
* Working memory complaints assessed by the Working Memory Questionnaire,
* Patients with a working memory disorder in at least one of the following tests: Digit Memory subtest WAIS-IV (standard deviation ≤ -2) , PASAT (percentile ≤ 10), Brown-Peterson (standard deviation ≤ -2).

Exclusion Criteria:

* Presence of aphasia, apraxia or severe neglect demonstrated by standardized neuropsychological tests during the inclusion visit: language - oral naming of BECS-GRECO images, ideational praxis and ideomotor , neglect - bell test,
* Insufficient visual or auditory abilities and oral and written expression to carry out neuropsychological tests,
* Severe depression assessed by the Beck Depression Inventory (BDI)
* Chronic alcoholic poisoning, drug addiction,
* Progressive general illness,
* Progressive psychiatric or neurological condition leading to cognitive impairment,
* Hospitalization for a neurological pathology since the acute phase of the qualifying event,
* Patient requiring surgery during study participation.
* Pregnant or breastfeeding women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Working memory performance | 8 weeks after baseline
  difference in performance on a working memory task (2-back) between phase A (therapeutic education) and interventional phase C (t-DCS + cognitive remediation) : a 2-back task is a repeated measure of working memory performance.
  On each trial, a stimulus will appear in the center of the screen for 500 msec. It will be followed by an inter-stimulus phase of 1500 msec. The stimulus will be a capital letter (consonants only). In this 2-back task, the subject will be asked to press the answer key as quickly as possible when the letter presented is identical to the penultimate. This task requires strong working memory and attentional resources. Error-free delay (ms), reaction times (ms) and standard deviation of reaction times (ms) will be counted.

SECONDARY OUTCOMES:
Goal attainment | 8 weeks after baseline
  The difference in Goal Attainment Scale (GAS) scores between phase A (therapeutic education) and interventional phase C (t-DCS + cognitive remediation).
  Each goal is personalized with the patient.
  The scale has 5 types of score each representing a goal attainment status (expectation) :
  * 2 being the further away form expectation
  * 1 a little less than aimed 0 meaning that the goal set is attained
    * 1 a little more than what was aimed
    * 2 exceeds a lot expectations

CONTACTS AND LOCATIONS:
Overall Officials: Adeline Julien, Principal Investigator — University Hospital, Toulouse